CLINICAL TRIAL: NCT04230824
Title: A Randomized, Double-blind, Placebo Controlled, Single-center Study to Determine the Effects of Pre-workout and Recovery Formulations on Soreness, Performance, Tolerance and Safety Outcomes in Healthy Adults Undergoing Training Program
Brief Title: Chronic Study on Body Composition, Training, Performance, and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20-PHX-0001 Chronic
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Damage Muscle; Body Weight Changes; Performance Enhancing Product Use
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-workout plus and Protein recovery plus (Active Comparator): Pre-workout plus: a blend of caffeine, choline bitartrate, carbohydrate, HMB, vitamin D3 mixed with water and consumed within 30 minutes prior to exercise
  Protein recovery plus: a blend of whey protein, caseinate, carbohydrate, vitamin C, alpha-tocopherol, vitamin D3, glucosamine mixed with water and consumed 15 minutes post exercise
  Interventions: Dietary Supplement: Pre-workout plus and Protein recovery plus; Other: 6-week resistance training program
- Placebo (Placebo Comparator): Non-caloric powder mixed with water and consumed within 30 minutes prior to exercise and within 15 minutes after exercise
  Interventions: Other: Placebo; Other: 6-week resistance training program
- Control (No Intervention): This arm will receive no intervention

INTERVENTIONS:
Dietary Supplement: Pre-workout plus and Protein recovery plus — products consumed prior and after exercise
  Arms: Pre-workout plus and Protein recovery plus
Other: Placebo — placebo product consumed prior and after exercise
  Arms: Placebo
Other: 6-week resistance training program — participants will complete a moderate-intensity warm-up, a full-body resistance training workout (2 x per week) and an interval training session (1 x per week)
  Arms: Placebo; Pre-workout plus and Protein recovery plus

SUMMARY:
The chronic phase of the study will evaluate the effects of pre-exercise and post-exercise ingestion of a multi-ingredient supplement on adaptations to a 6-week exercise program consisting of both resistance training and high intensity aerobic exercise, using a randomized, double-blind, placebo-controlled design. Participants will complete an enrollment/familiarization visit, a baseline testing session, followed by a 6-week supervised exercise intervention, and post-testing session identical to baseline testing. Participants will be randomized during the baseline session to groups receiving either 1) Active Treatment (pre-post supplementation), 2) placebo (noncaloric beverage), or 3) control, not participating in exercise or consuming a treatment. During the supervised 6-week resistance training program, participants will complete a moderate-intensity warm-up, a full-body resistance training workout (2 x per week) and an interval training session (1 x per week). Thirty-minutes prior to each training session, and within 15 minutes post-exercise, participants will consume their randomly assigned treatment beverage. Body composition, blood markers of muscle damage/recovery, strength, and performance tests will be measured before (baseline) and after training (Post) to evaluate the effects of supplementation. All data collection will be conducted by the Principal Investigator and Research Assistants. All subjects will report to the Applied Physiology Laboratory and Human Performance Center in Fetzer Hall for all testing and training sessions, which will span approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant is an adult between the ages of 25-50 years
* Participant has a recorded BMI of 20-35 kg/m2
* Participant exercises less than 3 hours per week for at least 8 weeks preceding the study
* Participant has provided written and dated informed consent to participate in the study
* Participant is willing to and able to comply with the protocol
* Participant is apparently healthy and no reported metabolic disorders, heart disease, arrhythmias, thyroid disease, renal, hepatic, autoimmune or neurological diseases, as determined by a health history questionnaire
* Participant agrees to maintain current diet and exercise routine during the study
* Participant agrees to refrain from taking any anti-inflammatory supplement 48 hours prior to exercise or for exercise related pain or medications to prevent any further nutritional or drug related protection against exercise induced muscle damage
* Participant agrees to wear an accelerometer to track activity during entire study
* Participant has a resting (seated for 5 minutes) blood pressure of systolic pressure between 140-90 mmHg and a diastolic pressure between 90-50 mmHg

Exclusion Criteria:

* Participant is currently enrolled in a separate clinical trial or weight loss program involving diet, exercise, physical activity, or the potential ingestion of an active drug or dietary supplement Participant is using, or has consistently used one of the following dietary supplements within 12 weeks prior to enrollment: Beta-alanine, Creatine, HMB, Carnosine, Vitamin D
* Participant has consistently consumed whey protein/plant protein and/or 1,000 mg of fish oil within the previous 4 weeks prior to enrollment
* Participant has gained or lost ≥ 8 lbs in the previous month
* Participant has a known allergy or sensitivity to the placebo or active ingredients
* Participant has used tobacco more than three days per week (on average) in the previous 6 months, or refuses to abstain from all tobacco use for the duration of the study
* Participant is pregnant or planning to become pregnant
* Participant has any musculoskeletal condition prohibiting them from participation

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Strength | baseline, week 8
  Change from baseline in strength by measuring 1 repetition maximum for leg press and bench press

SECONDARY OUTCOMES:
Muscle soreness | baseline, week 8
  Change from baseline on muscle soreness using visual analog scale (a horizontal 100 mm line where zero will represent no soreness and one-hundred will represent maximum amount of soreness. Participants will be asked to place a single vertical that represents their current soreness. The scale will be measured with a calibrated ruler with the higher numbers representing more soreness.)
Recovery | baseline, week 8
  Change from baseline on muscle damage by measuring creatine kinase and isoprostanes
Training Volume | baseline, week 8
  Change from baseline in total training volume measured by product of sets x repetitions completed x external load used in exercise routine
Performance | baseline, week 8
  Change from baseline on performance by measuring countermovement vertical jump
Body Composition | baseline, week 8
  Change from baseline in body composition using DXA measurements fat mass (kg) and lean mass (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabre HE, Gordon AN, Patterson ND, Smith-Ryan AE. Evaluation of pre-workout and recovery formulations on body composition and performance after a 6-week high-intensity training program. Front Nutr. 2022 Nov 2;9:1016310. doi: 10.3389/fnut.2022.1016310. eCollection 2022. PMID 36407519